CLINICAL TRIAL: NCT02595229
Title: Pronator Quadratus Repair After Volar Plating of Distal Radius Fractures or Not? - Results of a Prospective Randomized Trial
Brief Title: Pronator Quadratus Repair After Volar Plating of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2759/10
Record Dates: First submitted 2015-10-25; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Forearm Pronation Strength Recovery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PQ (Pronator quadraus) repair (Active Comparator): Following volar plate osteosynthesis the pronator quadratus muscle is sutured with 3 to 5 U-shaped stitches using a polyfilament absorbable synthetic suture.
  Interventions: Procedure: Pronator quadratus repair
- No PQ repair (No Intervention): Following volar plate osteosynthesis the pronator quadratus muscle is placed in its anatomical position without suture repair.

INTERVENTIONS:
Procedure: Pronator quadratus repair — Suturing of the pronator quadratus muscle
  Arms: PQ (Pronator quadraus) repair

SUMMARY:
Investigation of the influence of the pronator quadratus (PQ) muscle repair following volar plate fixation of distal radius fractures with regard to the forearm pronation strength. During the early recovery period of 3 months an improvement of pronation strength and functional scorings was hypothesized for the PQ repair when compared to no repair.

Randomization of the patients in two groups ( PQ repair and no repair) and follow-up examinations after 6 and 12 weeks included bilateral isometric pronation strength measurement, range of motion, the QuickDASH and the Mayo-Wrist-Score, and a visual analogue scale (VAS)

DETAILED DESCRIPTION:
Investigation of the influence of the pronator quadratus (PQ) muscle repair following volar plate fixation of distal radius fractures with special regards to the forearm pronation strength. During the early recovery period of 3 months an improvement of pronation strength and functional scorings was hypothesized for the PQ repair when compared to no repair.

Therefore the patients are randomized to group A = PQ repair and group B = no repair. Follow-up examinations after 6 and 12 weeks are scheduled included bilateral isometric pronation strength measurement, range of motion, the QuickDASH and the Mayo-Wrist-Score, and a visual analogue scale (VAS)

ELIGIBILITY:
Inclusion Criteria:

* isolated, closed fractures of the distal radius
* fractures type A2 to B2 according to the AO fracture classification system
* primary volar locking plate osteosynthesis within 7 days after trauma

Exclusion Criteria:

* concomitant fractures of the affected upper extremity
* intra-articular distal radius fractures ( type C)
* concomitant neurovascular injuries
* preexisting neurological illnesses
* initial external fixation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Isometric forearm pronation strength (N) | 6 weeks postoperative
  Measurement of the isometric forearm pronation strength (N) using the IsoForce-Control EVO 2 dynamometer (MDS AG, Oberburg, Switzerland)
Isometric forearm pronation strength (N) | 12 weeks postoperative
  Measurement of the isometric forearm pronation strength (N) using the IsoForce-Control EVO 2 dynamometer (MDS AG, Oberburg, Switzerland)

SECONDARY OUTCOMES:
Quick DASH Score (Patient-reported evaluation score for disabilities of the arm, shoulder and hand) | 6 weeks postoperative
  The score is assessed on the basis of a questionnaire (11 questions about disabilities in the daily life and symptoms as pain, sleeplessness, paresthesia)
Quick DASH Score (Patient-reported evaluation score for disabilities of the arm, shoulder and hand) | 12 weeks postoperative
  The score is assessed on the basis of a questionnaire (11 questions about disabilities in the daily life and symptoms as pain, sleeplessness, paresthesia)
Visual analogue scale (VAS) | 6 weeks postoperative
  Measurement of the pain level
Visual analogue scale (VAS) | 12 weeks postoperative
  Measurement of the pain level
Mayo-Wrist-Score (Physician-based evaluation score of the wrist function) | 6 weeks postoperative
  Assessment of the wrist function (grip strength, range of motion, pain intensity, functional status (return to work))
Mayo-Wrist-Score (Physician-based evaluation score of the wrist function) | 12 weeks postoperative
  Assessment of the wrist function (grip strength, range of motion, pain intensity, functional status (return to work))
Assessment of the bilateral wrist motion (AO neutral-0-method) | 6 weeks postoperative
  Measurement of the wrist motion using a goniometer, injured and uninjured hand (Pronation/ Supination, Ulnarabduction/ Radialabduction, Palmarflexion/ Dorsalextension)
Assessment of the bilateral wrist motion (AO neutral-0-method) | 12 weeks postoperative
  Measurement of the wrist motion using a goniometer, injured and uninjured hand (Pronation/ Supination, Ulnarabduction/ Radialabduction, Palmarflexion/ Dorsalextension)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Siebenlist, MD, Principal Investigator — Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Technische Universität München; Gunther Sandmann, MD, Principal Investigator — Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Technische Universität München

REFERENCES:
- [Derived] Haberle S, Sandmann GH, Deiler S, Kraus TM, Fensky F, Torsiglieri T, Rondak IC, Biberthaler P, Stockle U, Siebenlist S. Pronator quadratus repair after volar plating of distal radius fractures or not? Results of a prospective randomized trial. Eur J Med Res. 2015 Nov 25;20:93. doi: 10.1186/s40001-015-0187-4. PMID 26607745